CLINICAL TRIAL: NCT02376296
Title: Observational Study of Metastatic Prostate Cancer Subjects Receiving Docetaxel Therapy for Evaluation of Docetaxel Plasma Levels Using the MyDocetaxel Assay
Brief Title: Observational Study of Docetaxel Exposure in Metastatic Prostate Cancer Patients
Status: Completed | Type: Observational
Sponsor: Saladax Biomedical, Inc. (Industry)
Collaborators: UPMC CancerCenter (Unknown)
Responsible Party: Sponsor
Other Study IDs: SBI-DTX-004
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
Keywords: metastatic prostate cancer; castrate resistant prostate cancer; CRPC; hormone sensitive prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- hormone naïve: Subjects with hormone naïve metastatic prostate cancer that have high-volume disease and have been on androgen deprivation therapy for less than 120 days prior to starting docetaxel therapy.
  Interventions: Drug: docetaxel; Other: Blood draws
- castrate resistant: Subjects with castrate resistant prostate cancer (CRPC) [defined as having evidence of prostate specific antigen (PSA) progression despite androgen deprivation therapy] that have had at least four weeks elapse between the withdrawal of anti-androgens (Bicalutamide, Flutamide or Nilutamide) and the initiation of docetaxel therapy.
  Interventions: Drug: docetaxel; Other: Blood draws

INTERVENTIONS:
Drug: docetaxel — 3-weekly docetaxel therapy (starting dose of 75 mg/m2)
  Other Names: Taxotere
Other: Blood draws — Blood draws for determination of docetaxel plasma levels and exposure (AUC)

SUMMARY:
In this observational study, blood samples for pharmacokinetic (PK) testing will be collected from subjects with metastatic prostate cancer during their treatment with docetaxel. Plasma levels of docetaxel will be determined, and the subjects docetaxel exposure levels, determined as an area under the curve (AUC), will be retrospectively correlated with reports of toxicity, tumor response, quality of life, time to disease progression and overall survival to provide guidance on what the appropriate target range for docetaxel exposure should be for metastatic prostate cancer subjects receiving docetaxel therapy for their disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate.
* Male subjects 18 years of age or older.
* About to start a new line of treatment with docetaxel (75 mg/m2) in combination with prednisone.
* All subjects must be informed of the investigational nature of this study and be willing to provide written informed consent in accordance with Institutional guidelines and good clinical practices (GCP) indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study prior to the beginning of specific study procedures.
* Prior surgical castration or concurrent use of an agent for chemical castration with a serum testosterone level < 50 ng/dL.
* Subjects with hormone naïve metastatic prostate cancer, must have high-volume disease, defined as extra-nodal visceral disease or bone metastases with at least 4 bone lesions (one being outside of the vertebral column or pelvis).
* Subjects with hormone naïve high-volume metastatic prostate adenocarcinoma must have been on androgen deprivation therapy (including luteinizing hormone-releasing hormone (LHRH) agonist therapy, LHRH antagonist therapy, or surgical castration) for less than 120 days prior to starting docetaxel therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* For subjects with castrate resistant prostate cancer (CRPC), at least four weeks elapsed between withdrawal of anti-androgens (Bicalutamide, Flutamide or Nilutamide) and initiation of docetaxel therapy.
* For subjects with CRPC, at least four weeks elapsed between last administration of Abiraterone (Zytiga®) or Enzalutamide (Xtandi®) and initiation of docetaxel therapy.
* At least four weeks elapsed between prior surgery or prior radiotherapy and initiation of docetaxel therapy.
* Radiograph-documented evidence of soft tissue or bony metastatic disease.
* Must have adequate hematologic, hepatic and renal function as defined below:
* Hematologic (minimal values): Absolute neutrophil count ≥ 1,500/mm3; Hemoglobin ≥ 10.0 g/dl; Platelet count ≥ 75,000/mm3
* Hepatic Function: Total Bilirubin ≤ 1.5 x institutional upper limit of normal (ULN); asparate transaminase (AST) and alanine transaminase (ALT) < 2 x institutional ULN
* Suitable venous access and healthy enough (as determined by the treating physician) to provide whole blood sample.

Exclusion Criteria:

* Any condition / concomitant disease not allowing chemotherapy with docetaxel, prednisone or required premedication for the treatment regimen.
* Serious concurrent disorders (active infection requiring intravenous antibiotics, unstable angina, uncompensated congestive heart failure (CHF), or hepatic failure) that, in the opinion of the investigator, would prevent the use of docetaxel and/or compromise the subject's ability to provide whole blood samples for participation in the study.
* Concurrent use of any non-FDA approved (i.e. investigational or experimental) anticancer agent(s) or within four (4) weeks of enrolling on the study.
* Pre-existing neuropathy ≥ grade 2 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.
* Individuals with known seropositivity for human immunodeficiency virus (HIV), hepatitis C virus, hepatitis B surface antigen, or syphilis.
* Unwilling or unable to follow protocol requirements or to provide informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic prostate cancer patients, either newly diagnosed or castrate resistant, who are about to start treatment with a 3-weekly docetaxel treatment regimen (starting dose of 75 mg/m2) within the University of Pittsburgh Medical Center (UPMC) Cancer Center network.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-02; Primary Completion 2018-02-10 (Actual); Study Completion 2018-02-10 (Actual)

PRIMARY OUTCOMES:
Variability of docetaxel exposure | Up to 6 months after the initiation of docetaxel therapy
  Blood will be drawn during the first six cycles of docetaxel therapy to determine the variability of docetaxel exposure.
Docetaxel treatment related toxicities | Up to 7 months after the initiation of docetaxel therapy
  Determine the relationship between docetaxel plasma concentrations (i.e. exposure level) and the incidence of docetaxel related toxicities for identification of an optimal target docetaxel exposure range.

SECONDARY OUTCOMES:
Frequency of growth factor usage | Up to 7 months after the initiation of docetaxel therapy
  Determine relationship (if any) between growth factor usage and docetaxel exposure levels.
Number of days hospitalized for treatment of docetaxel related toxicities | Up to 7 months after the initiation of docetaxel therapy
  Determine relationship (if any) between number of day hospitalized due to treatment related toxicities and docetaxel exposure levels.
Time to prostate specific antigen (PSA) progression | Up to 24 months after the initiation of docetaxel therapy
  Determine relationship (if any) between the time to PSA progression and docetaxel exposure levels obtained during the first 6 cycles of treatment.
Tumor response as determined by imaging | Up to 7 months after the initiation of docetaxel therapy
  Determine relationship (if any) between the tumor response as determined by imaging and docetaxel exposure levels obtained during the first 6 cycles of treatment.
Changes in quality of life | Up to 6 months after the initiation of docetaxel therapy
  Determine relationship between changes in the quality of life (as measured using the FACT-P Questionnaire) and docetaxel exposure levels obtained during the first 6 cycles of treatment.
Overall survival | Up to 24 months after the initiation of docatexel therapy
  Determine relationship between overall survival and docetaxel exposure levels obtained during the first 6 cycles of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul A Parikh, MD, PhD, Principal Investigator — UPMC CancerCenter
Locations (20):
- United States (20):
  - UPMC CancerCenter - Beaver, Beaver, Pennsylvania
  - UPMC CancerCenter - Upper St. Clair, Bethel Park, Pennsylvania
  - UPMC CancerCenter - Horizon, Farrell, Pennsylvania
  - Arnold Palmer Cancer Center - Oakbrook, Greensburg, Pennsylvania
  - Arnold Palmer Cancer Center, Greensburg, Pennsylvania
  - UPMC CancerCenter - Greenville, Greenville, Pennsylvania
  - UPMC CancerCenter - Indiana, Indiana, Pennsylvania
  - UPMC CancerCenter at John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC CancerCenter - Mckeesport, McKeesport, Pennsylvania
  - UPMC CancerCenter - Monroeville, Monroeville, Pennsylvania
  - Arnold Palmer Medical Oncology - Mount Pleasant, Mount Pleasant, Pennsylvania
  - UPMC CancerCenter - New Castle, New Castle, Pennsylvania
  - UPMC CancerCenter - St. Margaret, Pittsburgh, Pennsylvania
  - UPMC CancerCenter - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC CancerCenter - Passavant HOA, Pittsburgh, Pennsylvania
  - UPMC CancerCenter - Passavant OHA, Pittsburgh, Pennsylvania
  - UPMC CancerCenter - Northwest, Seneca, Pennsylvania
  - UPMC CancerCenter - Uniontown, Uniontown, Pennsylvania
  - UPMC CancerCenter - Washington, Washington, Pennsylvania
  - UPMC CancerCenter - Jefferson, West Mifflin, Pennsylvania

IPD SHARING:
Plan to Share IPD: No